CLINICAL TRIAL: NCT01721798
Title: Comparison of Two Intrauterine Devices (IUDs) Among Cape Town HIV-positive Women: A Randomized Controlled Trial Assessing Safety of Registered Products in South Africa
Brief Title: Comparison of Two Intrauterine Devices (IUDs) Among Cape Town HIV-positive Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: University of Cape Town (Other); City University of New York, School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10369
Record Dates: First submitted 2012-10-18; First posted 2012-11-06 (Estimated); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-05

CONDITIONS: HIV
Keywords: AE adverse event; AIDS acquired immunodeficiency syndrome; ALT (SGPT) alanine aminotransferase; ART antiretroviral therapy; AST (SGOT) aspartate aminotransferase; DCF data collection forms; DMC Data Monitoring Committee; FDA (U.S.) Food and Drug Administration; GCP Good Clinical Practice guidelines; HB sAg Hepatitis B surface antigen; ICH International Council for Harmonization; IND Investigational New Drug Application; IRB Institutional Review Board; IU International units; mg milligram(s); mm3 cubic millimeter(s); PCR polymerase chain reaction; SAE serious adverse event; µg microgram; ULN upper limit of the normal range; WB Western Blot
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Copper T-380a Intrauterine Device (C-IUD) (Active Comparator): Copper T-380A Intrauterine Device with approximately 380 mm2 exposed copper. Devices used were those included as part of the South African public sector health formulary.
  Interventions: Device: Copper T-380a IUD
- Levonorgestrel IUD (LNG-IUD) (Active Comparator): Levonorgestrel IUD containing 52 mg levonorgestrel registered for contraceptive use in South Africa at the time of the trial.
  Interventions: Device: Mirena levonorgestrel IUD

INTERVENTIONS:
Device: Mirena levonorgestrel IUD — Intrauterine contraception system
  Arms: Levonorgestrel IUD (LNG-IUD)
Device: Copper T-380a IUD — intrauterine contraception system
  Arms: Copper T-380a Intrauterine Device (C-IUD)

SUMMARY:
This study will inform international medical guidelines as to whether the Levonorgestrel intrauterine device (LNG IUD), a highly effective long-acting reversible contraceptive method, is safe and acceptable as compared to the copper intrauterine device (C-IUD) for HIV-positive women in Cape Town, South Africa. If the LNG IUD is found to be safe and acceptable, the introduction of this method to HIV positive women in developing countries could significantly reduce unplanned pregnancy and mother-to-child transmission of HIV, and confer non-contraceptive benefits to HIV-positive women in Sub-Saharan Africa.

DETAILED DESCRIPTION:
Design: Single site, double-blind, randomized controlled trial

Population: HIV-positive South African women between the ages of 18 and 40 years

Study size: At least 166 women

Study intervention: Levonorgestrel intrauterine device (LNG IUD) or the copper T-380 intrauterine device (C-IUD)

Duration & Follow-up: Approximately 48 months in total. Recruitment will take approximately 24 months. After enrollment, each participant will be followed for 24 months.

Primary Objectives: To compare LNG IUD safety to the safety of the C-IUD with respect to genital HIV shedding, a surrogate for potential for HIV transmission, overall and in the presence and absence of antiretroviral therapy (ART).

Secondary Objectives: 1) To compare LNG IUD safety to the safety of the C-IUD with respect to HIV progression as measured by changes in plasma viral load (VL) at 6 months between the two pre-ART study arms. 2) To explore LNG IUD safety with respect to non-HIV related outcomes, including hemoglobin change, incidence of sexually-transmitted infections (STIs) and pelvic inflammatory disease (PID). 3) To measure LNG IUD acceptability through device continuation and other measures for the LNG IUD as compared to the C-IUD. 4) To compare three genital tract sampling methods to determine which provides optimal recovery of HIV RNA and immune mediators over a series of three visits.

Primary Endpoints: Change in detection and quantity of HIV ribonucleic acid (RNA) genital VL measures between study arms at baseline and 6 months, and over 24 months following IUD insertion.

Secondary Endpoints: 1) Measures of HIV disease progression, including CD4 change, time to ART initiation, and mean plasma VL change from baseline to 6 and through 24 months among pre-ART women. 2) Hemoglobin change and incidence of STIs and PID for all participants through 24 months. 3) IUD continuation and expulsion rates between study arms comparing different IUDs over a 24-month period and acceptability measures through quantitative and qualitative methods. 4) Comparison of female genital tract sampling methods for recovery of HIV RNA as measured by VL and immune mediators (e.g. cytokines).

Study Site: Gugulethu Community Health Centre (GCHC), Cape Town, South Africa

ELIGIBILITY:
Inclusion Criteria

* Willing and able to provide written informed consent (IC) to be screened for and to participate in the trial
* Interested and willing to use the intrauterine device (IUD) as a family planning method.
* Between 18 to 40 years of age (inclusive): This age range includes women during their years of greatest fertility and 18 is the age of majority for research consent in South Africa.
* Willing to participate in all aspects of the study and to comply with study procedures and visits, for 24 months, including:

  * Be randomized
  * Adhere to follow-up schedule and willing to be contacted by site staff between study visits (by phone and/or in person)
  * Provide contact/locator information
  * Agree for site staff to review clinic chart to confirm HIV status
* Has documented HIV infection
* For pre-antiretroviral therapy (ART) entrants:

  * ART-ineligible at screening, based on current South African ART guidelines
  * Be at least 6 months post-delivery and not pregnant or desiring pregnancy for the next 30 months.
* For ART-using entrants:

  * ART-use demonstrated by clinical records reflecting laboratory measures consistent with ART use and evidence of viral suppression (plasma viral load (VL)<1000 copies/mL) at the most recent VL measure.
  * Be at least 6 weeks post-delivery and not pregnant or desiring pregnancy for the next 30 months.
* Intending residence in Cape Town area for next 30 months
* No documented or known history of infertility or sterilization
* No gross evidence of cervical neoplasia on examination
* No prior history of ectopic pregnancy
* No history of or suspected hormonally-dependent neoplasm or undiagnosed abnormal vaginal bleeding
* Local language fluency and comprehension
* Not participating in any other clinical trial with a biomedical intervention
* Have no condition that, based on the opinion of the Site Principal Investigator (PI), would preclude provision of informed consent, make participation in the study unsafe, or complicate interpretation of data.

Exclusion Criteria:

* Known congenital or acquired uterine anomaly including fibroids distorting the uterine cavity;
* Known acute liver disease or hepatic neoplasm;
* Known copper storage disease;
* Known hypersensitivity to any component of the levonorgestrel IUD (LNG IUD) or copper IUD (C-IUD) or latex allergy
* Pregnant or desiring pregnancy in next 24 months
* Gross cervical lesion concerning for neoplasia
* CD4 lymphocyte count<350 cells/mm3 if not using ART
* Less than 6 weeks postpartum

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 199 (Actual)
Dates: Start 2013-11-10 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B Landon Myer, MBChB, PhD, Principal Investigator — University of Cape Town; Catherine Todd, MD, MPH, Principal Investigator — FHI 360
Locations (1):
- University of Cape Town, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Langwenya N, Todd CS, Jones HE, Hoover DR, Hu NC, Ronan A, Myer L. Risk-based screening to identify reproductive tract infection among HIV-infected women desiring use of intrauterine contraceptives. BMJ Sex Reprod Health. 2021 Apr;47(2):137-143. doi: 10.1136/bmjsrh-2019-200494. Epub 2020 Jul 1. PMID 32611546
- [Derived] Todd CS, Jones HE, Langwenya N, Hoover DR, Chen PL, Petro G, Myer L. Safety and continued use of the levonorgestrel intrauterine system as compared with the copper intrauterine device among women living with HIV in South Africa: A randomized controlled trial. PLoS Med. 2020 May 22;17(5):e1003110. doi: 10.1371/journal.pmed.1003110. eCollection 2020 May. PMID 32442189

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-ART/LNG-IUD: Not eligible to use antiretroviral therapy at enrollment (ART) at enrollment/ randomized to and received the levonorgestrel 52 mg intrauterine device (LNG-IUD)
- Non-ART/C-IUD: Not eligible to use antiretroviral therapy (ART) at enrollment/ randomized to and received the copper T380-A intrauterine device (C-IUD) containing approximately 380 mm2 of exposed copper surface area
- ART Use at Enrollment/LNG-IUD: Using antiretroviral therapy (ART) and virally suppressed (plasma viral load<1000 copies/mL) at enrollment/ randomized to and received the levonorgestrel 52 mg intrauterine device (LNG-IUD)
- ART Use at Enrollment/C-IUD: Using antiretroviral therapy (ART) and virally suppressed (plasma viral load<1000 copies/mL) at enrollment/ randomized to and received the copper T380-A intrauterine device (C-IUD) containing approximately 380 mm2 of exposed copper surface area
Period: Overall Study
Arm/Group | Non-ART/LNG-IUD | Non-ART/C-IUD | ART Use at Enrollment/LNG-IUD | ART Use at Enrollment/C-IUD
Started | 36 | 31 | 65 | 67
6 Mos | 35 | 30 | 60 | 62
12 Mos | 34 | 29 | 58 | 62
18 Mos | 32 | 29 | 55 | 60
Completed | 32 | 29 | 44 | 48
Not Completed | 4 | 2 | 21 | 19
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 2 | 2 | 9 | 9
Not completed — Pregnancy | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 1
Not completed — Not eligible for 24 month visit | 1 | 0 | 8 | 7

BASELINE CHARACTERISTICS:
Population: Women of reproductive age living with HIV
Groups:
- Non-ART/LNG-IUD: Not using ART at Enrollment (per national guidelines at study start, ART eligibility was initially limited to CD4<350 cells/mm3. This criteria was changed in 2015 to a threshold of CD4<500 cells/mm3 with an accompanying protocol amendment and then again in 2016 when ART initiation at diagnosis became standard of care, with a further protocol amendment. As such, there are relatively few participants in this arm.)/ LNG-IUD (the hormonal IUD used in this study is a T-shaped device containing 52mg levonorgestrel, releasing 20 mcg levonorgestrel daily.)
- Non-ART/C-IUD: Not using ART at Enrollment: (per national guidelines at study start, ART eligibility was initially limited to CD4<350 cells/mm3. This criteria was changed in 2015 to a threshold of CD4<500 cells/mm3 with an accompanying protocol amendment and then again in 2016 when ART initiation at diagnosis became standard of care, with a further protocol amendment. As such, there are relatively few participants in this arm.) /C-IUD (The copper IUD used in this study is the copper T Cu380A, containing 380 mm2 of exposed copper wire.)
- ART Use at Enrollment/LNG-IUD: Using ART at Enrollment (two new study arms were added in 2015 to include women using ART with clinical viral suppression (plasma viral load<1000 copies/mL) and change the primary outcome measure to detectable genital HIV RNA)/LNG-IUD (the hormonal IUD used in this study is a T-shaped device containing 52mg levonorgestrel, releasing 20 mcg levonorgestrel daily.)
- ART Use at Enrollment/C-IUD: Using ART at Enrollment (two new study arms were added in 2015 to include women using ART with clinical viral suppression (plasma viral load<1000 copies/mL) and change the primary outcome measure to detectable genital HIV RNA)/C-IUD (The copper IUD used in this study is the copper T Cu380A, containing 380 mm2 of exposed copper wire.)
- Total: Total of all reporting groups
Arm/Group | Non-ART/LNG-IUD | Non-ART/C-IUD | ART Use at Enrollment/LNG-IUD | ART Use at Enrollment/C-IUD | Total
Number analyzed (Participants) | 36 | 31 | 65 | 67 | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 36 | 31 | 65 | 67 | 199
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.6 (4.6) | 30.2 (5.0) | 31.8 (4.5) | 32.1 (4.8) | 31.4 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 31 | 65 | 67 | 199
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 36 | 31 | 65 | 67 | 199
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 36 | 31 | 65 | 67 | 199
Recent (<=16 weeks) exposure to injectable progestin contraception [Count of Participants; unit: Participants] | 15 | 12 | 25 | 26 | 78

OUTCOME MEASURES:

1. Primary Outcome: Participants With Detectable Genital Tract HIV Ribonucleic Acid (RNA) Viral Load (VL)
Description: Number of women with detectable genital tract HIV RNA as measured with menstrual cup sampling at each scheduled visit. Level of detection was 20-40 copies/mL depending on assay; outcome was dichotomous with copies above level of detection coded as detectable and those below level of detection considered undetectable.
Time Frame: Enrollment to 24 months
Population: As-treated contributing any person-time at follow-up; proportions with detectable genital tract HIV RNA compared in longitudinal analysis.
Measure: Number; unit: Participants
Groups:
- Non-ART (Not Using Antiretroviral Therapy)/ Levonorgestrel Intrauterine Device (LNG-IUD): Not eligible to use antiretroviral therapy (ART) at enrollment/ randomized to and received the levonorgestrel 52 mg intrauterine device (LNG-IUD)
Arm/Group | Non-ART (Not Using Antiretroviral Therapy)/ Levonorgestrel Intrauterine Device (LNG-IUD) | Non-ART/C-IUD | ART Use at Enrollment/LNG-IUD | ART Use at Enrollment/C-IUD
Number analyzed (Participants) | 36 | 31 | 65 | 67
Participants
  Enrollment | 18 | 23 | 10 | 7
  3 mos: number analyzed (Participants) | 36 | 27 | 60 | 64
  3 mos | 19 | 18 | 8 | 11
  6 mos: number analyzed (Participants) | 35 | 29 | 60 | 62
  6 mos | 20 | 14 | 11 | 15
  12 mos: number analyzed (Participants) | 34 | 29 | 58 | 62
  12 mos | 21 | 16 | 5 | 10
  18 mos: number analyzed (Participants) | 32 | 28 | 55 | 60
  18 mos | 22 | 13 | 11 | 14
  24 mos: number analyzed (Participants) | 32 | 29 | 44 | 48
  24 mos | 14 | 10 | 8 | 13
Statistical Analysis 1: Comparison: Non-ART (Not Using Antiretroviral Therapy)/ Levonorgestrel Intrauterine Device (LNG-IUD) vs Non-ART/C-IUD vs ART Use at Enrollment/LNG-IUD vs ART Use at Enrollment/C-IUD; C-IUD is comparator group; Test type: Non-Inferiority — Primary Outcome Analysis: Proportion of women with detectable genital viral load across 24 months; p = 0.66, GEE; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.47 to 1.62]

2. Secondary Outcome: Participants With Detectable Plasma HIV Ribonucleic Acid (RNA) Viral Load Among Those Using Antiretroviral Therapy (ART)
Description: The proportion of women using ART at enrollment with detectable plasma HIV RNA viral load. Viral load assays detected HIV RNA levels at 20-40 copies/mL as the lower limit of detection. The outcome measure coded values above that limit as detectable and those below as undetectable for women using ART and in mean viral load for women not using ART.
Time Frame: Enrollment to 24 months
Population: Women recorded as using ART at a scheduled study visit with continued use of allocated intrauterine device.
Measure: Number; unit: Participants
Arm/Group | ART Use at Enrollment/LNG-IUD | ART Use at Enrollment/C-IUD
Number analyzed (Participants) | 65 | 67
Participants
  Enrollment: number analyzed (Participants) | 65 | 64
  Enrollment | 14 | 12
  3 mos: number analyzed (Participants) | 60 | 62
  3 mos | 11 | 20
  6 mos: number analyzed (Participants) | 60 | 62
  6 mos | 18 | 19
  12 mos: number analyzed (Participants) | 58 | 55
  12 mos | 18 | 22
  18 mos: number analyzed (Participants) | 55 | 56
  18 mos | 15 | 20
  24 mos: number analyzed (Participants) | 44 | 44
  24 mos | 14 | 21
Statistical Analysis 1: Comparison: ART Use at Enrollment/LNG-IUD; C-IUD is comparator group; Test type: Non-Inferiority — Secondary Outcome Analysis of Proportion with Detectable plasma viral load users at 24 months; p = 0.64, GEE; Adjusted as-treated analysis; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.37 to 1.86]

3. Secondary Outcome: Mean Hemoglobin Concentration as Part of Intrauterine Contraceptive Safety
Description: Participant hemoglobin measured at baseline, 6, 12, 18, and 24 months with blood sample with mean hemoglobin calculated and trends over time assessed. Other safety measures were included with this secondary outcome, such as adverse events, summarized with descriptive statistics.
Time Frame: Enrollment to 24 months
Population: Participants continuing use of the allocated intrauterine device (IUD) and having hemoglobin measured at 6-month intervals.
Measure: Mean (Standard Deviation); unit: grams/deciliter
Groups:
- Non-antiretroviral Therapy (ART)/ Levonorgestrel Intrauterine Device (LNG-IUD): Not eligible to use antiretroviral therapy (ART) at enrollment/ randomized to and received the levonorgestrel 52 mg intrauterine device (LNG-IUD)
- Non-antiretroviral Therapy (ART)/ Copper T380A Intrauterine Device (C-IUD): Not eligible to use antiretroviral therapy (ART) at enrollment/ randomized to and received the copper T380-A intrauterine device (C-IUD) containing approximately 380 mm2 of exposed copper surface area
Arm/Group | Non-antiretroviral Therapy (ART)/ Levonorgestrel Intrauterine Device (LNG-IUD) | Non-antiretroviral Therapy (ART)/ Copper T380A Intrauterine Device (C-IUD) | ART Use at Enrollment/LNG-IUD | ART Use at Enrollment/C-IUD
Number analyzed (Participants) | 36 | 31 | 65 | 67
grams/deciliter
  Enrollment | 12.4 (1.3) | 12.8 (1.0) | 12.4 (1.1) | 12.2 (1.3)
  6 months: number analyzed (Participants) | 35 | 29 | 60 | 62
  6 months | 12.6 (1.3) | 12.3 (1.2) | 12.5 (1.4) | 11.8 (1.6)
  12 months: number analyzed (Participants) | 34 | 29 | 58 | 62
  12 months | 12.5 (1.1) | 12.3 (0.89) | 12.6 (0.86) | 11.8 (1.4)
  18 months: number analyzed (Participants) | 32 | 28 | 55 | 60
  18 months | 12.4 (1.0) | 12.4 (0.85) | 12.6 (1.4) | 11.7 (1.3)
  24 months: number analyzed (Participants) | 32 | 29 | 44 | 48
  24 months | 12.6 (1.0) | 12.6 (1.7) | 12.6 (0.91) | 11.6 (1.1)

4. Secondary Outcome: Participants Continuing Use of the Allocated Intrauterine Device (IUD)
Description: Measure of the number of women continuing to use the allocated intrauterine device (IUD) across all visits as a measure of acceptability. Proportion of women using the allocated IUD measured at each scheduled visit with time using the IUD adjusted for discontinuation at unscheduled visits. Continuation rate analyzed longitudinally with Kaplan-Meier survival analysis.
Time Frame: Enrollment to 24 months
Population: Participants receiving the allocated IUD and contributing follow-up time at scheduled and unscheduled (e.g., request for IUD removal) visits. Analysis was proportion of women continuing their allocated IUD over time. The denominator at each scheduled visit changed based on number presenting or eligible (at 24 mos) for follow-up visits.
Measure: Number; unit: Participants
Groups:
- Non-ART/Copper T380A Intrauterine Device (C-IUD): Not eligible to use antiretroviral therapy (ART) at enrollment/ randomized to and received the copper T380-A intrauterine device (C-IUD) containing approximately 380 mm2 of exposed copper surface area
- ART/LNG-IUD: Using antiretroviral therapy (ART) and virally suppressed (plasma viral load<1000 copies/mL) at enrollment/ randomized to and received the levonorgestrel 52 mg intrauterine device (LNG-IUD)
- ART/C-IUD: Using antiretroviral therapy (ART) and virally suppressed (plasma viral load<1000 copies/mL) at enrollment/ randomized to and received the copper T380-A intrauterine device (C-IUD) containing approximately 380 mm2 of exposed copper surface area
Arm/Group | Non-antiretroviral Therapy (ART)/ Levonorgestrel Intrauterine Device (LNG-IUD) | Non-ART/Copper T380A Intrauterine Device (C-IUD) | ART/LNG-IUD | ART/C-IUD
Number analyzed (Participants) | 36 | 31 | 65 | 67
Participants
  Enrollment | 36 | 31 | 65 | 67
  3 mos: number analyzed (Participants) | 36 | 24 | 60 | 61
  3 mos | 36 | 21 | 60 | 58
  6 mos: number analyzed (Participants) | 35 | 25 | 60 | 58
  6 mos | 35 | 20 | 60 | 49
  12 mos: number analyzed (Participants) | 34 | 23 | 57 | 51
  12 mos | 33 | 18 | 56 | 39
  18 mos: number analyzed (Participants) | 30 | 22 | 51 | 43
  18 mos | 28 | 16 | 49 | 31
  24 mos: number analyzed (Participants) | 30 | 18 | 41 | 33
  24 mos | 28 | 13 | 38 | 23
Statistical Analysis 1: Comparison: Non-ART/Copper T380A Intrauterine Device (C-IUD) vs ART/C-IUD; C-IUD is comparator group; Test type: Non-Inferiority — Secondary Outcome Analysis of Allocated IUC continuation at 24 months; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 8.61, 95% CI 2-sided [3.03 to 24.4]

5. Secondary Outcome: HIV Ribonucleic Acid (RNA) Concentration by Lower Female Genital Tract Sampling Method
Description: Proportion of specimens with quantifiable genital viral load compared by specific sampling method (menstrual cup, endocervical swab, and swab-enriched lavage) at enrollment, 3 months and 6 months among women not using antiretroviral therapy (ART). Allocated intrauterine device (IUD) was not considered in this analysis.
Time Frame: 6 months
Population: Women living with HIV who were not using ART receiving the allocated intrauterine device (IUD) had lower genital tract samples taken for genital tract viral load by three different methods: menstrual cup, endocervical swab, & swab-enriched lavage, at enrollment, 3-, and 6-month visits. Sampling order varied by visit (e.g., enrollment: menstrual cup, endocervical swab, endocervical swab-enriched lavage). The number in each group was different at enrollment, 3 months and 6 months.
Measure: Count of Participants; unit: Participants
Groups:
- Menstrual Cup: Genital tract samples from enrollment, three, and six-month visits for women not using antiretroviral therapy (ART) allocated to either levonorgestrel intrauterine device (LNG-IUD) or copper intrauterine device (C-IUD).
- Swab-enriched Lavage: Female lower genital tract samples obtained through rotated flocked endocervical swab followed by lavage with 1.5 mL of phosphate buffered saline. Swab tips were stored with recovered lavage fluid.
- Endocervical Swab: Genital tract samples obtained through flocked swab rotated in the endocervical canal.
Arm/Group | Menstrual Cup | Swab-enriched Lavage | Endocervical Swab
Number analyzed (Participants) | 51 | 51 | 51
Participants
  Enrollment: number analyzed (Participants) | 47 | 48 | 51
  Enrollment | 28 | 18 | 21
  3 months: number analyzed (Participants) | 46 | 48 | 48
  3 months | 26 | 14 | 21
  6 months: number analyzed (Participants) | 43 | 49 | 49
  6 months | 19 | 16 | 23

ADVERSE EVENTS:
Time Frame: Participant follow-up time was up to 24 months; we followed unresolved adverse events a further 3-6 months until a final disposition was recorded.
Groups:
- Non-ART/LNG-IUD: Not using ART at Enrollment/LNG-IUD
- Non-ART/C-IUD: Not using ART at Enrollment//C-IUD
- ART Use at Enrollment/LNG-IUD: Using ART at Enrollment/LNG-IUD
- ART Use at Enrollment/C-IUD: Using ART at Enrollment/C-IUD
- All Women Using LNG-IUD: All women with equal to or more than one event using LNG-IUD
- All Women Using C-IUD: All women with equal to or more than one event using C-IUD
Arm/Group | Non-ART/LNG-IUD | Non-ART/C-IUD | ART Use at Enrollment/LNG-IUD | ART Use at Enrollment/C-IUD | All Women Using LNG-IUD | All Women Using C-IUD
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/31 | 1/65 | 1/67 | 1/101 | 1/98
Serious Adverse Events (participants affected / at risk) | 12/36 | 12/31 | 8/65 | 7/67 | 20/101 | 19/98
Other Adverse Events (participants affected / at risk) | 36/36 | 31/31 | 63/65 | 65/67 | 99/101 | 96/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-ART/LNG-IUD (N=36) | Non-ART/C-IUD (N=31) | ART Use at Enrollment/LNG-IUD (N=65) | ART Use at Enrollment/C-IUD (N=67) | All Women Using LNG-IUD (N=101) | All Women Using C-IUD (N=98)
Depression (Psychiatric disorders) | 0 | 3 | 0 | 0 | 0 | 3
Low CD4 count (Immune system disorders) | 9 | 5 | 0 | 0 | 9 | 5 — In keeping with the South Africa's 2015 guideline for initiation of ART based on CD4<=500, participant's CD4 count necessitated ART referral under new clinical guidelines.
Gallstones (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 1 | 0
Pelvic Inflammatory Disease (Reproductive system and breast disorders) | 1 | 1 | 2 | 0 | 3 | 1
Pregnancy with IUD in place (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 0 | 1 | 1
Mood disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hernia Surgery (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Death - possibly injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Liver failure/injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Car accident- Broken Leg - Hospitalization (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Accident - Broken Leg - Hospitalization (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Abscess/Vagina Labia Majora (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Right Tubal Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 1
Admission to psychiatric hospital (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cervical intraepithelial neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Death - unknown reasons (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
IUD expulsion (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-ART/LNG-IUD (N=36) | Non-ART/C-IUD (N=31) | ART Use at Enrollment/LNG-IUD (N=65) | ART Use at Enrollment/C-IUD (N=67) | All Women Using LNG-IUD (N=101) | All Women Using C-IUD (N=98)
Amenorrhea (Blood and lymphatic system disorders) | 17 | 3 | 32 | 8 | 49 | 11
Menorrhagia (Blood and lymphatic system disorders) | 2 | 11 | 3 | 17 | 5 | 28
Intermenstrual bleeding (Blood and lymphatic system disorders) | 10 | 5 | 13 | 17 | 23 | 22
Irregular/heavy uterine bleeding (Blood and lymphatic system disorders) | 4 | 6 | 4 | 7 | 8 | 13
Menstrual disorder (Blood and lymphatic system disorders) | 0 | 0 | 7 | 5 | 7 | 5
Pelvic pain (Reproductive system and breast disorders) | 17 | 15 | 12 | 15 | 29 | 30
Dysmenorrhea (Reproductive system and breast disorders) | 3 | 8 | 3 | 7 | 6 | 15
Enlarged Abdomen (Reproductive system and breast disorders) | 3 | 2 | 3 | 5 | 6 | 7
Breast Pain (Reproductive system and breast disorders) | 0 | 1 | 3 | 6 | 3 | 7
Lower back pain (Reproductive system and breast disorders) | 4 | 2 | 1 | 0 | 5 | 2
Leukorrhea (Infections and infestations) | 2 | 4 | 3 | 6 | 5 | 10
Cervicitis (Infections and infestations) | 2 | 1 | 3 | 0 | 2 | 1
Weight gain (General disorders) | 5 | 5 | 6 | 8 | 11 | 13
Weight loss (General disorders) | 0 | 0 | 2 | 1 | 2 | 1
Headache (General disorders) | 7 | 3 | 2 | 4 | 9 | 7
Anaemia (Blood and lymphatic system disorders) | 2 | 8 | 1 | 2 | 3 | 10
Nausea (General disorders) | 2 | 5 | 5 | 1 | 7 | 6
Acne (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT01721798/Prot_SAP_000.pdf
  • Informed Consent Form (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT01721798/ICF_001.pdf